CLINICAL TRIAL: NCT06049004
Title: Investigation of the Validity and Reliability of the Londrina Activities of Daily Living Protocol in Idiopathic Pulmonary Fibrosis Patients
Brief Title: Londrina Activities of Daily Living Protocol in Idiopathic Pulmonary Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof., Izmir Katip Celebi University
Other Study IDs: IKC124
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Activity, Motor
Keywords: idiopathic pulmonary fibrosis; activity daily living; validity; reliability
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Activities of Daily Living Protocol — The protocol is a performance-based objective measurement method based on repetition of daily activities. Participants are asked to perform the activities defined in the protocol at the same speed they do at home. The Londrina Protocol includes 5 stations: Station 1 Arranging Objects on the Table, Station 2 Walking with Bags, Station 3 Organizing Shelves, Station 4 Clothesline Task, Station 5 Walking. The completion time of the protocol is recorded.

SUMMARY:
The Londrina Activities of Daily Living Protocol was first developed for Chronic Obstructive Pulmonary Disease patients and was found to be valid and reliable, but there is no validity and reliability study of the Londrina Activities of Daily Living Protocol in IPF patients. The purpose of the study is to Examine the Validity and Reliability of the Londrina Activities of Daily Living Protocol in Idiopathic Pulmonary Fibrosis (IPF) patients.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is an interstitial lung disease characterized by a restrictive type of breathing disorder. In IPF patients, serious limitations occur in the activities of daily living (ADL) of the patients due to dyspnea and fatigue symptoms, therefore it is very important to evaluate the activities of daily living in this patient group. It is recommended to use protocols created from activities frequently used in daily life to evaluate ADL in chronic respiratory patients. Londrina Activities of Daily Living Protocol is a performance-based objective measurement method based on repetition of daily activities. Participants are asked to perform the activities defined in the protocol at the same speed they do at home, and the completion time of the protocol is recorded. The individual is asked to complete all stations in order from a designated starting line.

The Londrina Activities of Daily Living Protocol was first developed for Chronic Obstructive Pulmonary Disease patients and was found to be valid and reliable, but there is no validity and reliability study of the Londrina Activities of Daily Living Protocol in IPF patients. The purpose of our study is to Examine the Validity and Reliability of the Londrina Activities of Daily Living Protocol in IPF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with idiopathic pulmonary fibrosis (IPF) disease
2. Being 18 years or older
3. Being independent in daily living activities
4. Being able to read and understand Turkish

Exclusion Criteria:

1. The patient refuses to participate in the study
2. People with comorbidities that would make it impossible to perform any of the study evaluations (orthopedic pathology, uncontrolled cardiovascular or neurological conditions, psychiatric illness, etc.)
3. Presence of infection in the last 3 months
4. Those who show changes in their usual symptoms during the protocol
5. Patients who have difficulty understanding the commands given
6. Those who cannot complete all evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being diagnosed with idiopathic pulmonary fibrosis (IPF) disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Londrina Activities of Daily Living Protocol | 15 minutes
  The protocol is a performance-based objective measurement method based on repetition of daily activities. Participants are asked to perform the activities defined in the protocol at the same speed they do at home. The Londrina Protocol includes 5 stations: Station 1 Arranging Objects on the Table, Station 2 Walking with Bags, Station 3 Organizing Shelves, Station 4 Clothesline Task, Station 5 Walking. The completion time of the protocol is recorded.

SECONDARY OUTCOMES:
Glittre Activities of Daily Living Test: | 5 minutes
  The test is a submaximal exercise test developed by selecting activities similar to activities of daily living to evaluate functional capacity in COPD. The test provides information about performance in activities of daily living and may reflect functional capacity. It is a test that takes place within a distance of 10 m in total. During the test, female patients carry a 2.5 kg backpack and male patients carry a 5 kg backpack. The test involves five rounds and patients are asked to complete these rounds as quickly as possible. Test completion time is recorded. Glittre ADL Test is a valid and reliable test in patients with idiopathic pulmonary fibrosis.
London Chest Activities of Daily Living (ADL) Scale | 10 minutes
  Used in diseases such as COPD and heart failure, to evaluate dyspnea that occurs only with activities of daily living, Garrod et al. It is a simple, standardized, valid and reliable questionnaire developed by . This survey consists of 4 parts. It consists of 15 items in total: self-care: 4 items, housework 6 items, physical activity 2 items, and leisure activities 3 items. Each item is given a score ranging from 0 to 5. The total score varies between 0-75. Higher scores indicate greater ADL limitations.
Hand Grip Strength Measurement | 5 minutes
  A hand dynamometer will be used to evaluate grip strength (Lafayette Professional Hand Dynamometer 5030L1, USA). Participants were placed in the standard test position determined by the American Association of Hand Therapists for grip strength measurement.
mMRC Dyspnea Scale | 5 minutes
  This scale is a five-item scale (0: no dyspnea, 4 severe dyspnea) based on various physical activities that cause the feeling of dyspnea. Here, patients are asked to mark the level of activity that causes dyspnea.
Respiratory Function Test | 10 minutes
  Measurements will be made with a portable spirometer device. Forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), percentages of the FEV1/FVC ratio according to expected values according to age, height, body weight and gender, and inspiratory and expiratory respiratory muscle forces will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No